CLINICAL TRIAL: NCT03371030
Title: Role of the Pronator Quadratus in Vascularity and Stabilisation in Distal Radius Fractures After Osteosynthesis: Clinical and Anatomical Experimental Study
Brief Title: Role of the Pronator Quadratus in Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-QUA-2017-36
Record Dates: First submitted 2017-11-29; First posted 2017-12-13 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Radius; Fracture, Lower or Distal End
Keywords: distal radius fractures; pronator quadratus; osteosynthesis
MeSH Terms: conditions — Fractures, Bone; Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pronator quadratus reparation (Experimental): Surgical Intervention: Radius fracture teated with plate and pronator quadratus muscle repair.
  Interventions: Procedure: Pronatus quadratus reparation
- No pronator quadratus reparation (Active Comparator): Surgical Intervention: Radius fracture with plate without pronator quadratus muscle repair.
  Interventions: Procedure: Pronatus quadratus reparation

INTERVENTIONS:
Procedure: Pronatus quadratus reparation — Displaced and intra-articular distal radius fractures treated with volar approach and plate fixation. Pronator Quadratus muscle repair.

SUMMARY:
The skin, the bones, and most muscles received branches from the source arteries of at least two angiosomes, thus revealing one of the important anastomotic pathways by which the circulation is reconstituted in those cases where a source artery is interrupted by disease or trauma.

There are numerous metaphyseal-epiphyseal branches arise within the pronator quadratus and the anterior interosseous artery and course towards the distal radius. These branches may be fundamental to the healing of the distal radius fractures and make nonunion a rare complication. The aim of this study is the evaluation of the role of the pronator quadratus muscle and its repair in volar approach in distal radius fractures treated with plate fixation.

DETAILED DESCRIPTION:
Nonunion is an extremely rare complication in distal radius fractures and is most likely to occur in patients with conditions such as diabetes, peripheral vascular disease, or alcoholism. Diagnosis of nonunion is based on the absence of radiographic signs of union at 6 months. Treatment should be individualized but options are reconstructive procedures or wrist arthrodesis. In volar plating and often by the fracture injury itself, the complete pronator quadratus is stripped off the volar radius. Thus, the intraosseous collateral circulation must be sufficient for clinical healing. Any operative approach to the distal radius fracture should not compromise both volar radial and the dorsoulnar arteries.

While the branches to the pronator quadratus must be sacrificed in a palmar approach, the distal perforator can and should be spared. This is true even in the flexor carpi radialis extended approach. In distal radius fractures, when the normal outward flow of blood through the cortex is blocked, the periosteal arterioles have more ability than medullary arterioles to function and proliferate.

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fractures with intra-articular fragment, comminuted or displaced fracture
* Adults between 18- 90 years old

Exclusion Criteria:

* Children
* Non displaced distal radius fractures treated with immobilization.
* Adults older than 90 years old

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Fracture consolidation | 3 months
  X-Ray radius union

SECONDARY OUTCOMES:
Clinical stability | 3 months
  Clinical stability of the distal radioulnar joint
Radiological stability | 3 months
  Radiological stability of the distal radioulnar joint

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lamas, MD, Ph D, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haerle M, Schaller HE, Mathoulin C. Vascular anatomy of the palmar surfaces of the distal radius and ulna: its relevance to pedicled bone grafts at the distal palmar forearm. J Hand Surg Br. 2003 Apr;28(2):131-6. doi: 10.1016/s0266-7681(02)00279-6. PMID 12631484
- [Background] Inoue Y, Taylor GI. The angiosomes of the forearm: anatomic study and clinical implications. Plast Reconstr Surg. 1996 Aug;98(2):195-210. doi: 10.1097/00006534-199608000-00001. PMID 8764707
- [Background] Orbay J, Badia A, Khoury RK, Gonzalez E, Indriago I. Volar fixed-angle fixation of distal radius fractures: the DVR plate. Tech Hand Up Extrem Surg. 2004 Sep;8(3):142-8. doi: 10.1097/01.bth.0000126570.82826.0a. PMID 16518106
- [Background] Sheetz KK, Bishop AT, Berger RA. The arterial blood supply of the distal radius and ulna and its potential use in vascularized pedicled bone grafts. J Hand Surg Am. 1995 Nov;20(6):902-14. doi: 10.1016/S0363-5023(05)80136-4. PMID 8583061
- [Background] Huang HK, Wang JP, Chang MC. Repair of Pronator Quadratus With Partial Muscle Split and Distal Transfer for Volar Plating of Distal Radius Fractures. J Hand Surg Am. 2017 Nov;42(11):935.e1-935.e5. doi: 10.1016/j.jhsa.2017.08.018. PMID 29101976
- [Background] Lamas C, Llusa M, Mendez A, Proubasta I, Carrera A, Forcada P. Intraosseous vascularity of the distal radius: anatomy and clinical implications in distal radius fractures. Hand (N Y). 2009 Dec;4(4):418-23. doi: 10.1007/s11552-009-9204-9. Epub 2009 May 28. PMID 19475457
- [Derived] Lamas C, Arenas J, Almenara M, Rojas R, Fa-Binefa M, Toro-Aguilera A. Is pronator quadratus muscle repair required after anterior plate fixation for distal radial fractures? A prospective randomized comparative study. J Hand Surg Eur Vol. 2024 Mar;49(3):334-340. doi: 10.1177/17531934231192337. Epub 2023 Sep 8. PMID 37684023